CLINICAL TRIAL: NCT02221687
Title: Evaluation of the Efficacy and Safety of an Infant Formula Containing Synbiotics and Its Effects on the Incidence of Infectious Diseases in the Infant Gut : a Double-blind, Randomized, Controlled Interventional Study
Brief Title: The Combiotic-Study
Acronym: GOLFIII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment of breastfed infants was very slow. Decision with PI (05/2018): Termination (80/100); no implication on primary outcome. Predetermined number of breastfed infants (n=100) was arbitray choice. Formula groups completed (460/460) 12/2017.
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 505564 - PEC10561
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Healthy Term Infants
Keywords: synbiotic formula; infant formula; diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Synbiotic formula (Experimental): Synbiotic formula : standard formula enriched with a prebiotic fiber and a probiotic strain
  Dose : variable number of powder scoops, adapted to the infant's age and weight, and addition of the defined amount of water, according to the Dose and Drinking Amount table.
  Route : oral, ad libitum
  Duration of product intake:
  * Synbiotic IF : 5 months of consumption (from the inclusion until 6 months completed of age)
  * Synbiotic FoF: 6 months of consumption (from 6 to 12 months of age)
  Interventions: Dietary Supplement: Synbiotic formula
- Control formula (Placebo Comparator): Control formula : standard formula without pre and probiotic
  Dose : variable number of powder scoops, adapted to the infant's age and weight, and addition of the defined amount of water according to the Dose and Drinking Amount table.
  Route: oral, ad libitum
  Duration of product intake:
  * Control IF : 5 months of consumption (from the inclusion until 6 months completed of age)
  * Control FoF : 6 months of consumption (from 6 to 12 months of age)
  Interventions: Dietary Supplement: Control formula
- Breast-fed group (No Intervention): - Breast milk as exclusive feeding (no more than one formula meal per day), from birth until at least 4 months of age. Then, when the mother decides to stop breastfeeding, the infants can consume any formula on parent's choice respecting forbidden products list.
  Dose:
  * Breast milk : on demand
  Route : oral, ad libitum
  Duration of product intake:
  * Breast milk : at least 4 month (from birth until at least 4 months of age)

INTERVENTIONS:
Dietary Supplement: Synbiotic formula — Standard milk formula enriched with a prebiotic fiber and a probiotic strain
  Arms: Synbiotic formula
Dietary Supplement: Control formula — Standard milk formula without pre and probiotic
  Arms: Control formula

SUMMARY:
The primary objective of this study is to demonstrate that a synbiotic formula, fed for the duration of the first year of life (infant and follow-on formula) reduces the incidence rate of episodes of infectious diarrhea in infants during the first year of life compared to a standard infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants
* Female or male gender
* Gestational age between 37 and 41 weeks completed (= 41 weeks + 6 days)
* Age at time of V1 visit : 4 +/- 7 days
* Birth weight between 2500 ans 4200g, with regular weight gain (≥ 150g / week)
* Two legal representatives (parent(s) / guardian(s)) who are capable of and willing to comply with the protocol and have signed the informed consent in accordance with legal requirements.
* at least one of the legal representatives is affiliated to with a social security scheme.

Additionnaly , criteria of inclusion in one of the formula-fed groups or in the breast-fed group, respectively, are the following:

* To be included in one of the formula arm, infants will have to be exclusively formula-fed (no breast milk meal) at the time of V1 visit (randomization).

or

* To be included in the breastfeeding arm, infants will have to be exclusively breast-fed (no more than one formula meal per day) at V1 visit (randomization) and its mother will have to be willing to pursue exclusive breastfeeding at least until the infant will be 4-month old.

Exclusion Criteria:

* Intensive care during at least the first 14 days of life
* Neonatal health problems, such as: respiratory distress, asphyxia, hypoglycemia, sepsis, NEC (necrotizing enterocolitis),...
* Clinical evidence of chronic illness or gastrointestinal disorders such as : GER (Gastrooesophageal Reflux), gastroenteritis,...
* Known metabolic disorders, such as diabetes, lactose intolerance,....
* Known immune deficiency
* Subjects recommended to receive formula with hydrolized protein (e.g. children with allergy risk)
* Subject under oral antibiotic treatment at V1 visit
* Participation in another biomedical study
* Whose legal representatives have psychological or linguistic incapability to sign the informed consent form
* Reasons to presume that parents are unable to meet the study plan requirements (e.g. impossibility to contact study representatives in case of emergency, drug addiction etc)

Ages: 3 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
(Cumulative) number of infectious diarrhea episodes per subject during the first year of life. | one year
  Difference between formula groups are evaluated via incidence rate based on number of subjects.
  In formula-fed infants, diarrhea is defined as three or more loose or watery stools in 24 hours with or without fever or vomiting (according to WHO and ESPGHAN definition). For breast-fed infants, a change in stool consistency versus previous stool consistency is more indicative of diarrhea than stool number.
  Diarrhea episode is considered as ended as soon as 2 consecutive non-watery stools are observed or no stools are observed in 24 hours.

SECONDARY OUTCOMES:
Analysis of fecal microbiota by molecular analysis from frozen stools in planned stool samples | 4 months
  Levels of total lactobacilli, Lactobacillus fermentum species (and if possible the strain CECT 5716 will be quantified too), total bifidobacteria, enterobacteriaceae, clostridium difficile
Analysis of fecal microbiota by molecular analysis from frozen stools in planned stool samples | 1 year
  Levels of total lactobacilli, Lactobacillus fermentum species (and if possible the strain CECT 5716 will be quantified too), total bifidobacteria, enterobacteriaceae, clostridium difficile
Analysis of fecal microbiota by molecular analysis from frozen stools in planned stool samples | 2 years
  Levels of total lactobacilli, Lactobacillus fermentum species (and if possible the strain CECT 5716 will be quantified too), total bifidobacteria, enterobacteriaceae, clostridium difficile
Analysis of fecal microbiota by molecular analysis from frozen stools in planned stool samples | 3 years
  Levels of total lactobacilli, Lactobacillus fermentum species (and if possible the strain CECT 5716 will be quantified too), total bifidobacteria, enterobacteriaceae, clostridium difficile
Analysis of fecal microbiota by molecular analysis from frozen stools in diarrhea samples | 1 year
  levels of potential pathogens causing diarrhea including rotavirus, norovirus, Salmonella enterica, Campylobacter jejuni, Clostridium difficile, Clostridium perfringens, Escherichia coli (potential pathogenic bacteria will be screened only in case of negative testing for viruses on sample collected within 72 hours after beginning of the diarrhea episode);
Fecal pH and levels of short chain fatty acids (SCFA) in planned stool samples | 4 months
  short chain fatty acids (SCFA): acetate, propionate, butyrate;
Fecal pH and levels of short chain fatty acids (SCFA) in planned stool samples | 1 year
  short chain fatty acids (SCFA): acetate, propionate, butyrate;
Fecal pH and levels of short chain fatty acids (SCFA) in planned stool samples | 2 years
  short chain fatty acids (SCFA): acetate, propionate, butyrate;
Fecal pH and levels of short chain fatty acids (SCFA) in planned stool samples | 3 years
  short chain fatty acids (SCFA): acetate, propionate, butyrate;
Characteristics of bowel movements and stools | 4 months
  - assessed through a 3-day diary filled in by parents
  * average daily number of bowel movements;
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) (using the validated scale for preterm and term infants proposed by Bekkali N, et al., 2009), and especially
  * average daily incidence of loose or watery stools (category A, subscale 'consistency' on Bekkali scale);
  * dominant stool color per visit
Characteristics of bowel movements and stools | 6 months
  - assessed through a 3-day diary filled in by parents
  * average daily number of bowel movements;
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) (using the validated scale for preterm and term infants proposed by Bekkali N, et al., 2009), and especially
  * average daily incidence of loose or watery stools (category A, subscale 'consistency' on Bekkali scale);
  * dominant stool color per visit
Characteristics of bowel movements and stools | 9 months
  - assessed through a 3-day diary filled in by parents
  * average daily number of bowel movements;
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) (using the validated scale for preterm and term infants proposed by Bekkali N, et al., 2009), and especially
  * average daily incidence of loose or watery stools (category A, subscale 'consistency' on Bekkali scale);
  * dominant stool color per visit
Characteristics of bowel movements and stools | 1 year
  - assessed through a 3-day diary filled in by parents
  * average daily number of bowel movements;
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) (using the validated scale for preterm and term infants proposed by Bekkali N, et al., 2009), and especially
  * average daily incidence of loose or watery stools (category A, subscale 'consistency' on Bekkali scale);
  * dominant stool color per visit
Characteristics of bowel movements and stools | 2 years
  - assessed through a 3-day diary filled in by parents
  * average daily number of bowel movements;
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) (using the validated scale for preterm and term infants proposed by Bekkali N, et al., 2009), and especially
  * average daily incidence of loose or watery stools (category A, subscale 'consistency' on Bekkali scale);
  * dominant stool color per visit
Characteristics of bowel movements and stools | 3 years
  - assessed through a 3-day diary filled in by parents
  * average daily number of bowel movements;
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) (using the validated scale for preterm and term infants proposed by Bekkali N, et al., 2009), and especially
  * average daily incidence of loose or watery stools (category A, subscale 'consistency' on Bekkali scale);
  * dominant stool color per visit
Characteristics of bowel movements during diarrhea episodes | 1 year
  - assessed through a diary filled in by parents during diarrhea episodes
  * average daily number of bowel movements per diarrhea episode;
  * average duration (number of days) of diarrhea episodes;
  * total number of days with diarrhea, within the first year of age (between V1 and V5);
  * (average daily) Infant Stool Form scores consistency (4-point scale), amount (4-point scale) and color (6 categories) per diarrhea episode.
Levels of fecal IgA and fecal calprotectin in planned stool samples | 4 months
Levels of fecal IgA and fecal calprotectin in planned stool samples | 1 year
Levels of fecal IgA and fecal calprotectin in planned stool samples | 2 years
Levels of fecal IgA and fecal calprotectin in planned stool samples | 3 years
Number and duration of infectious diseases | 3 years
  Especially: otitis media, infections of upper and lower respiratory tract and of urinary tract;
Number and duration of fever episodes; | 3 years
Number and duration of antibiotic treatment. | 3 years
Infants growth measured by anthropometric measurements | 4 weeks
  weight, size, head circumference;
Infants growth measured by anthropometric measurements | 4 months
  weight, size, head circumference;
Infants growth measured by anthropometric measurements | 6 months
  weight, size, head circumference;
Infants growth measured by anthropometric measurements | 9 months
  weight, size, head circumference;
Infants growth measured by anthropometric measurements | 1 year
  weight, size, head circumference;
Infants growth measured by anthropometric measurements | 2 years
  weight, size, head circumference;
Infants growth measured by anthropometric measurements | 3 years
  weight, size, head circumference;
Child's behavior | 4 months
  Assessed through a 3-day diary filled in by parents
  - Average sleep duration and crying duration per 24 hours;
Child's behavior | 6 months
  Assessed through a 3-day diary filled in by parents
  - Average sleep duration and crying duration per 24 hours;
Child's behavior | 9 months
  Assessed through a 3-day diary filled in by parents
  - Average sleep duration and crying duration per 24 hours;
Child's behavior | 1 year
  Assessed through a 3-day diary filled in by parents
  - Average sleep duration and crying duration per 24 hours;
Child's behavior | 2 years
  Assessed through a 3-day diary filled in by parents
  - Average sleep duration and crying duration per 24 hours;
Child's behavior | 3 years
  Assessed through a 3-day diary filled in by parents
  - Average sleep duration and crying duration per 24 hours;
Minor gastrointestinal disorders (digestive tolerance) | 4 months
  Assessed through a 3-day diary filled in by parents
  - average daily vomiting, regurgitation/reflux, flatulence, constipation (according to WHO definition);
Minor gastrointestinal disorders (digestive tolerance) | 6 months
  Assessed through a 3-day diary filled in by parents
  - average daily vomiting, regurgitation/reflux, flatulence, constipation (according to WHO definition);
Minor gastrointestinal disorders (digestive tolerance) | 9 months
  Assessed through a 3-day diary filled in by parents
  - average daily vomiting, regurgitation/reflux, flatulence, constipation (according to WHO definition);
Minor gastrointestinal disorders (digestive tolerance) | 1 year
  Assessed through a 3-day diary filled in by parents
  - average daily vomiting, regurgitation/reflux, flatulence, constipation (according to WHO definition);
Minor gastrointestinal disorders (digestive tolerance) | 2 years
  Assessed through a 3-day diary filled in by parents
  - average daily vomiting, regurgitation/reflux, flatulence, constipation (according to WHO definition);
Minor gastrointestinal disorders (digestive tolerance) | 3 years
  Assessed through a 3-day diary filled in by parents
  - average daily vomiting, regurgitation/reflux, flatulence, constipation (according to WHO definition);
Suitability for daily use | 4 months
  Assessed through a 3-day diary filled in by parents
  - average daily consumption: drinking amounts and formula acceptance;
Suitability for daily use | 6 months
  Assessed through a 3-day diary filled in by parents
  - average daily consumption: drinking amounts and formula acceptance;
Suitability for daily use | 9 months
  Assessed through a 3-day diary filled in by parents
  - average daily consumption: drinking amounts and formula acceptance;
Suitability for daily use | 1 year
  Assessed through a 3-day diary filled in by parents
  - average daily consumption: drinking amounts and formula acceptance;
Suitability for daily use | 2 years
  Assessed through a 3-day diary filled in by parents
  - average daily consumption: drinking amounts and formula acceptance;
Suitability for daily use | 3 years
  Assessed through a 3-day diary filled in by parents
  - average daily consumption: drinking amounts and formula acceptance;
Adverse events (AE) | 4 months
  Assessed through a 3-day diary filled in by parents
  - Number of events, number of subjects showing adverse events, intensity and relationship of AE.
Adverse events (AE) | 6 months
  Assessed through a 3-day diary filled in by parents
  - Number of events, number of subjects showing adverse events, intensity and relationship of AE.
Adverse events (AE) | 9 months
  Assessed through a 3-day diary filled in by parents
  - Number of events, number of subjects showing adverse events, intensity and relationship of AE.
Adverse events (AE) | 1 year
  Assessed through a 3-day diary filled in by parents
  - Number of events, number of subjects showing adverse events, intensity and relationship of AE.
Adverse events (AE) | 2 years
  Assessed through a 3-day diary filled in by parents
  - Number of events, number of subjects showing adverse events, intensity and relationship of AE.
Adverse events (AE) | 3 years
  Assessed through a 3-day diary filled in by parents
  - Number of events, number of subjects showing adverse events, intensity and relationship of AE.
Number and duration of fever episodes; | 1 year
Number and duration of antibiotic treatment. | 1 year
Number and duration of infectious diseases | 1 year
  Especially: otitis media, infections of upper and lower respiratory tract and of urinary tract;

OTHER OUTCOMES:
Microbiota results | 1 year
  Phyla and families of bacteria in planned stools using 16S taxonomical metasequencing compared to the control formula in a sub-group of 96 infants only
Urinary D-Lactate and creatinine | 4 weeks
  To assess change in the urinary lactate and creatinine (in a subgroup of 96 infants only) via ratio after 3 months of consumption of the supplemented infant formula, compared to the control formula
Urinary D-Lactate and creatinine | 4 months
  To assess change in the urinary lactate and creatinine (in a subgroup of 96 infants only) via ratio after 3 months of consumption of the supplemented infant formula, compared to the control formula
Microbiota results | 4 months
  Phyla and families of bacteria in planned stools using 16S taxonomical metasequencing compared to the control formula in a sub-group of 96 infants only
Microbiota results | 2 years
  Phyla and families of bacteria in planned stools using 16S taxonomical metasequencing compared to the control formula in a sub-group of 96 infants only
Microbiota results | 3 years
  Phyla and families of bacteria in planned stools using 16S taxonomical metasequencing compared to the control formula in a sub-group of 96 infants only

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Piloquet, Pediatrician, Principal Investigator
Locations (25):
- France (25):
  - Elie JABBOUR, Gémozac, Charente-Maritime
  - Christophe VIEL, La Rochelle, Charente-Maritime
  - C.I.C Pédiatrique - C.H.U. de Grenoble - Hôpital Couple-Enfant, Grenoble, Isère
  - C.I.C pédiatrique - C.H.U. de Nantes - Hôpital Mère-Enfant, Nantes, Loire-Atlantique
  - Alain PALOMBA, Angers, Maine-et-Loire
  - Christophe RONDEAU, Angers, Maine-et-Loire
  - Damien GODIN, Angers, Maine-et-Loire
  - Daniel GOMBAUD, Angers, Maine-et-Loire
  - Jean-François FOUCAULT, Angers, Maine-et-Loire
  - Michel LAMBERT, Angers, Maine-et-Loire
  - Nolwenn RONCERAY, Angers, Maine-et-Loire
  - Philippe REMAUD, Angers, Maine-et-Loire
  - Pierre-André FERRAND, Angers, Maine-et-Loire
  - Vanessa BERNAND, Angers, Maine-et-Loire
  - Francisco MARTINEZ-CORTES, Angers, Maine-et-Loire
  - Damien GUILLON, Angers, Maine-et-Loire
  - Christine REGIMBART, Bécon-les-Granits, Maine-et-Loire
  - Antoine LEPELLETIER, Montreuil, Maine-et-Loire
  - Benoit DAGUZAN, Segré, Maine-et-Loire
  - Didier NOURRY, Tiercé, Maine-et-Loire
  - Philippe IGIGABEL, Tiercé, Maine-et-Loire
  - Alain BATY, Laval, Mayenne
  - Christian DUROY, Laval, Mayenne
  - François RICHARD, Laval, Mayenne
  - Patrick ROBERT, Laval, Mayenne

REFERENCES:
- [Derived] Piloquet H, Vrignaud B, Gillaizeau F, Capronnier O, Berding K, Gunther J, Hecht C, Regimbart C; GOLF III Study Group. Efficacy and safety of a synbiotic infant formula for the prevention of respiratory and gastrointestinal infections: a randomized controlled trial. Am J Clin Nutr. 2024 May;119(5):1259-1269. doi: 10.1016/j.ajcnut.2024.03.005. Epub 2024 Mar 10. PMID 38462218
- [Derived] Lagkouvardos I, Intze E, Schaubeck M, Rooney JP, Hecht C, Piloquet H, Clavel T. Early life gut microbiota profiles linked to synbiotic formula effects: a randomized clinical trial in European infants. Am J Clin Nutr. 2023 Feb;117(2):326-339. doi: 10.1016/j.ajcnut.2022.11.012. Epub 2022 Dec 21. PMID 36811568